CLINICAL TRIAL: NCT04860050
Title: A Double Blind, Parallel, Placebo-controlled, Randomised Clinical Trial to Evaluate the Efficacy of Turmipure Gold® to Improve Cognitive Performance in Healthy Aging.
Brief Title: Turmeric for Memory Impairment and Cognition
Acronym: TURMEMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-125
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Change; Mood; Stress
Keywords: Turmeric; Curcuminoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPG (Experimental): 76 participants who meet the eligibility criteria will be randomized under experimental arm and will receive Turmipure GOLD® product during 24 weeks
  Interventions: Dietary Supplement: Turmipure Gold®
- Control (Placebo Comparator): 76 participants who meet the eligibility criteria will be randomized under experimental arm and will receive placebo (colored acacia gum) product during 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Turmipure Gold® — TPG: Turmipure GOLD® - 1 capsule per day - as prescribed
  Arms: TPG
Dietary Supplement: Placebo — Placebo: colored acacia gum - 1 capsule per day - as prescribed
  Arms: Control

SUMMARY:
The objective of the study is to test the capacity of acute and chronic supplementations of Turmipure GOLD® to improve cognitive performance in healthy aging

DETAILED DESCRIPTION:
The aim of this clinical study is to determine whether oral administration of Turmipure GOLD® can contribute to the short- and long-term improvement of cognitive functions, including memory and attention, in subjects with age-associated memory impairment.

ELIGIBILITY:
Inclusion Criteria:

* Consent to the study and willing/able to comply with study product
* Males and females aged ≥ 60 and ≤ 85 years old
* Participants with subjective memory impairment, with preserved global cognitive functions, everyday activities, and no dementia, fulfilling age-associated memory impairment criteria based on the following National Institute of Mental Health criteria (AAMI, Crook 1986):

  1. Subjective memory complaint reflected in everyday difficulties (gradual) confirmed with a MAC-Q ≥25
  2. Memory loss confirmed by a 1st degree relative or life-partner
  3. Memory test performance that is at least 1SD below the mean established for healthy adults on a standardised test of secondary memory (VPA I and II portions of the Wechsler Memory Scale IV)
  4. Evidence of adequate intellectual function as determined by the Vocabulary subset of the Wechsler Adult Intelligence Scale
  5. Absence of dementia, as determined by the Telephone - Mini-Mental State Examination (MMSE) predicted in person score ≥24
* Not suffering from depression or anxiety, as determined by the Hospital Anxiety and Depression Scale (HADs) score of ≤7 for both depression and anxiety
* With a BMI between 18 and 32 kg/m²
* With a glycated haemoglobin/A1C score ≤ 5.7 %
* Willing to maintain existing dietary, body weight, and physical activity patterns throughout the study period

Exclusion Criteria:

* Abnormal laboratory test results of clinical significance
* With significant cardiovascular history, or significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude supplement ingestion and/or assessment of safety and the study objectives, as deemed exclusionary by the Principal Investigator
* With history of major head trauma, chronic traumatic encephalopathy, epilepsy, cerebrovascular disease, stroke or clinically diagnosed with mild cognitive impairment or dementia (such as Alzheimer's Disease according to the NINCDS-ADRDA guidelines), acute psychiatric disorder, schizophrenia, mania, depression (within past 24 months) or under any concurrent medical, cognitive or psychiatric condition that would either: compromise his/her ability to comply with the study requirements, may pose significant risk to the subject, or be deemed exclusionary by the Principal Investigator
* History of heavy smoking (> 1 pack/day) within past 3 months
* History of heavy caffeinated beverage consumption (> 400 mg caffeine/day) within past 2 weeks
* Taking any supplements or vitamins notably known to affect cognitive function (e.g. Living Nutrition Cognitive, Viridian Cognitive Complex, fish oil etc., list not exhaustive), or any psychotropic medications and products which interact with acetylcholine esterase and/or NMDA receptors (6-week washout before screening). Vitamin D and Calcium supplements permitted if on a stable dose for the previous 3 months
* Participant with history of drug and/or alcohol abuse at the time of enrolment
* Significant change of dietary habits within the preceding month
* With known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon or significant systemic disease, and with history of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years
* Participant with known allergy to components of the test product or with a medical history of food allergies
* Having uncontrolled hypertension, uncontrolled hypothyroidism or hyperthyroidism or uncontrolled lipidaemia (hypercholesteremia or hypertriglyceridemia) that is not on stable medication for at least 3 months.
* Current illnesses which could interfere with the study (e.g. prolonged severe diarrhoea, regurgitation/severe, difficulty swallowing)
* Participants taking any anticoagulant (including aspirin) or heparin treatment
* Participant currently involved in any other clinical trial or having participated in a trial within the preceding 90 days
* Individuals who are unable to give informed consent
* Participant has a history of non-compliance with medical treatments or recommendations
* Occupations that resulted in disruption of sleep-wake cycles
* Participant has difficulty hearing with or without a hearing aid or is colour blind or is visually impaired

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance through Quality of Working memory | 24 weeks
  Quality of Working memory is a composite score determined by the CDR System™ test battery (unit: #)

SECONDARY OUTCOMES:
Change in cognitive performance through Power of Attention | 24 weeks
  Power of Attention is a composite score determined by the CDR System™ test battery (unit: ms)
Change in cognitive performance through Continuity of Attention | 24 weeks
  Continuity of Attention is a composite score determined by the CDR System™ test battery (unit: #)
Change in cognitive performance through Cognitive Reaction Time | 24 weeks
  Cognitive Reaction Time is a composite score determined by the CDR System™ test battery (unit: ms)
Change in cognitive performance through Speed of Memory | 24 weeks
  Speed of Memory is a composite score determined by the CDR System™ test battery (unit: ms)
Change in cognitive performance through Quality of Episodic Memory | 24 weeks
  Quality of Episodic Memory is a composite score determined by the CDR System™ test battery (unit: #)
Change in cognitive performance through Quality of Memory | 24 weeks
  Quality of Memory is a composite score determined by the CDR System™ test battery (unit: #)
Change in cognitive performance through Executive Function | 24 weeks
  Executive Function is a composite score determined by the CDR System™ test battery (unit: #)
Change in stress | 24 weeks
  Stress will be assessed using the validated scale Perceived Stress Scale (0 to 56, higher scores meaning at maximum stress)
Change in feelings and emotions | 24 weeks
  Mood will be assessed using the validated Positive and Negative Affect Schedule - Expanded Form (PANAS-X) questionnaire
Change in mood | 24 weeks
  Mood will be assessed using the validated Bond-Lader questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Professor, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided